CLINICAL TRIAL: NCT00680303
Title: The Effect of Spacing of Lidcombe Program Clinic Visits
Brief Title: Spacing Lidcombe Program Clinic Visits
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sydney (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Newcastle University (Other)
Responsible Party: Professor Mark Onslow, Australian Stuttering Research Centre, The University of Sydney
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 402763-17; 402763
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-04

CONDITIONS: Stuttering
Keywords: Early Stuttering; Lidcombe Program; Stuttering Treatment; Efficiency; Efficacy; Service Delivery; Models of intervention
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): The child will receive the Lidcombe Program 2x per week
  Interventions: Behavioral: The Lidcombe Program for early stuttering
- 2 (Experimental): The child will receive the Lidcombe Program once every 2 weeks (fortnightly visits)
  Interventions: Behavioral: The Lidcombe Program for early stuttering
- 3 (Other): The child will receive the standard Lidcombe Program once per week (control)
  Interventions: Behavioral: The Lidcombe Program for early stuttering

INTERVENTIONS:
Behavioral: The Lidcombe Program for early stuttering
  Arms: 2
Behavioral: The Lidcombe Program for early stuttering
  Arms: 3
Behavioral: The Lidcombe Program for early stuttering
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the efficiency of the Lidcombe Program for early stuttering by varying the time between clinic visits during the first stage of the program.

DETAILED DESCRIPTION:
Stuttering is a communicative disorder that affects an estimated 5.19% of children. Although approximately 71.4% of children whose stuttering onset is in the preschool years exhibit spontaneous recovery within two years after first reported onset, there remain a significant number of children who require fluency intervention. Given the potential for negative long term social and communicative consequences due to persistent stuttering, there is a consensus among speech-language pathologists that stuttering should be treated early. However, the longer a child's stuttering persists, the less likely the child will spontaneously recover.

The Lidcombe Program is a behavioral therapy program for preschool children designed to treat stuttering at its early stages. The treatment approach involves the direct participation of parents, who are trained during parent and child weekly visits to a speech language pathologist. In the first stage of the program, the clinician demonstrates the therapy to the parent, observes the parent conduct therapy and provides feedback and goals for the following week until the next clinic visit. The clinician guides the parent to provide three types of verbal "reinforcement" contingencies for the child's stutter free speech. These include, acknowledgment, praise and request for self-evaluation, where the child is asked to recognize his or her stutter free speech. If unambiguous stuttering occurs, the parent provides two types of verbal "punishment" contingencies including acknowledgment of the stuttering and request for self-correction, where the child is asked to repeat the stuttered word again. These contingencies are administered by parents in everyday speaking conversations, in order to promote generalization of fluent speech. When the child's stuttering is reduced to near-zero levels, the child then enters the second stage of the program, where the number of clinic visits are gradually phased out from bi-monthly to monthly to every 2 months, and so on, as required by the child. The purpose of the stage 2 visits is for the speech language pathologist to evaluate the child's speech and to ensure that near-zero stuttering levels are maintained.

When the first stage of the Lidcombe program is followed as the program was originally designed, the median treatment time to achieve the criteria of near-zero levels of stuttering is 11 one-hour weekly clinic visits, with treatment times varying according to the severity of the stuttering. However, clinicians have been deviating from the standard weekly sessions for various reasons. For instance, some private practitioners are offering first stage treatment visits once every 2 weeks rather than weekly and other practitioners are offering treatment intensively, so that clients from remote areas can have access to the Lidcombe program. As yet, there are no data to confirm whether treatment using fortnightly or twice weekly clinic visits is as effective or efficient as the standard weekly visits. The aim of this project is to evaluate the following questions: (1) Does altering the spacing of LP clinic visits affect treatment efficiency? (2) Does altering the spacing of LP clinic visits affect treatment efficacy?

ELIGIBILITY:
Inclusion Criteria:

1. 3;0-5;11 years of age
2. Stuttering for longer than 6 months
3. Functional English spoken by parent and child
4. Stuttering over 2%SS in one Beyond Clinic measure
5. Diagnosis of stuttering

Exclusion Criteria:

1. Less than 2%SS
2. Previous treatment for stuttering in last 6 months
3. Parental report of ADHD or intellectual disability

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
1. Number of clinic visits required to achieve Stage II (0-1%SS, Severity Rating=1) 2. Number of clinic days to achieve Stage II 3. Percent Syllables Stuttered (%SS) at entry to Stage II | Entry into Stage II

SECONDARY OUTCOMES:
Parent reported Severity Ratings (SR) | Pre-treatment, entry into Stage 2, 9 months post-randomization, 18 months post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Mark Onslow, Principal Investigator — University of Sydney
Locations (2):
- University of Newcastle, Newcastle, New South Wales, Australia
- The Montreal Fluency Centre, Montreal, Quebec, Canada